CLINICAL TRIAL: NCT02591160
Title: Optimal Hydrochlorothiazide Cessation in Diagnosis of Hyperparathyroidism
Brief Title: Optimal HCTZ Cessation for Diagnosis of Hyperparathyroidism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Robert P. Zitsch III, William E Davis Professor and Chair, University of Missouri-Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1213821
Record Dates: First submitted 2015-10-27; First posted 2015-10-29 (Estimated); Last update posted 2018-01-08 (Actual); Status verified 2018-01

CONDITIONS: Hyperparathyroidism
MeSH Terms: conditions — Hyperparathyroidism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HCTZ cessation (Other): Patients will stop taking HCTZ for 3 months while submitting serial blood and 24 hour urine samples
  Interventions: Procedure: HCTZ cessation

INTERVENTIONS:
Procedure: HCTZ cessation — Patients will stop taking their HCTZ for 3 months

SUMMARY:
Primary hyperparathyroidism (PHPT) is the most common cause of hypercalcemia in the ambulatory setting. PHPT may be cured with surgery and indications for intervention have been defined and include urinary calcium/creatinine clearance. Hydrochlorothiazide (HCTZ), the most commonly prescribed medication for hypertension, reduces urinary calcium excretion and confounds urinary testing. As a result, it is universally recommended that thiazide diuretics be stopped in advance of urinary testing. To date, no studies are available to provide evidence-based guidance as to how long HCTZ must be held for urinary calcium excretion to return to steady state in PHPT. The objective of this study is to serially calculate urinary calcium/creatinine clearance ration in patients with suspected PHPT while holding HCTZ to determine the minimum duration of medication cessation necessary for urinary calcium clearance to reach steady state.

DETAILED DESCRIPTION:
In this study, adult patients will submit serum and 24 hour urine samples prior to HCTZ cessation and at the following intervals after cessation: 4-6 days, 14-16 days, 28-30 days, adn 90-92 days. To minimize confounding variable, patients will take supplemental Vitamin D and Calcium, monitor their daily calcium intake, and monitor blood pressure weekly. Alternative, non-diuretic, antihypertensive medication(s) may be prescribed at the discretion of the enrolling provider.

ELIGIBILITY:
Inclusion Criteria:

1. Elevated calcium on at least two separate draws with coexistent elevated parathyroid hormone (PTH) on at least one occasion.
2. Taking Hydrochlorothiazide for hypertension
3. Following a "wash period", patients must have a normal range 25-hydroxy Vitamin D level, thyroid stimulation hormone (TSH) and serum magnesium levels.
4. Controlled blood pressure
5. Willingness to comply with serial sampling
6. English as the primary language
7. Adults 18 years and older

Exclusion Criteria:

1. Unable to cease Hydrochlorothiazide for any reason
2. Congestive heart failure
3. Renal insufficiency (GFR <60)
4. Cardiovascular event in the last 3 months - include myocardial infarction, new onset atrial fibrillation, and new onset bundle branch block
5. Take lithium or other diuretic medication in last 3 months
6. Positive family history of familial hypocalciuric hypercalcemia (FHH)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2017-09-13 (Actual); Study Completion 2017-09-13 (Actual)

PRIMARY OUTCOMES:
Number of days for Calcium/Creatinine Clearance to normalize after stopping HCTZ | 2-3 years
  Determination of the HCTZ cessation window

CONTACTS AND LOCATIONS:
Overall Officials: Robert P Zitsch, MD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared.